CLINICAL TRIAL: NCT06922916
Title: Perioperative Risk Factors Related to the Prognosis of Lung Transplantation: A Retrospective Study
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chair of the Department of Anesthesiology, Zhejiang University
Other Study IDs: ZJU2025B0268
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: COPD; Interstitial Pneumonia; Bronchiectasis; Respiratory Failure; Idiopathic Pulmonary Fibrosis (IPF); Silicosis; Pulmonary Tuberculosis; Pulmonary Hypertension; Pulmonary Heart Disease
Keywords: lung transplantatipn; Perioperative-related risks; Mortality; In-hospital complications; Prognosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Bronchiectasis; Respiratory Insufficiency; Idiopathic Pulmonary Fibrosis; Silicosis; Tuberculosis, Pulmonary; Hypertension, Pulmonary; Pulmonary Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lung transplantation group: In this group, we collected perioperative clinical data and analyzed risk factors associated with patient outcomes.

SUMMARY:
This study analyzes patients who underwent lung transplantation at the First Affiliated Hospital of Zhejiang University from 2017 to 2024, focusing on anesthesia's impact on post-op results. It gathers patient data from hospital and Mediston systems, with main focus on in-hospital complications and secondary focus on ICU stay, post-op hospitalization, mortality, and intubation time. The research aims to deepen understanding of anesthetic management's role in lung transplant outcomes and guide improvements in perioperative anesthesia protocols.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years at time of transplantation
* Received single or bilateral lung transplantation

Exclusion Criteria:

* Re-transplantation
* Multi-organ transplantation
* Autotransplantation
* Incomplete medical records: Recipients with >20% missing essential data elements in any of these categories:Preoperative baseline characteristics； Intraoperative parameters；Postoperative outcome measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent lung transplantation at the First Affiliated Hospital of Zhejiang University between January 2017 and October 2024
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-04-22 (Estimated); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
In-hospital adverse events | Collect data for an expected average about 2 hours
  In-hospital adverse events were defined as post-transplant complications occurring prior to discharge, such as: Grade 3 PGD, respiratory infections, stroke, cardiac events, AKI, or liver impairment.

SECONDARY OUTCOMES:
ICU stay | Collect data for an expected average about 2 hours
  The ICU stay （days） was calculated from the time of ICU admission after surgery completion to actual discharge from the intensive care unit
Postoperative hospital stay | Collect data for an expected average about 2 hours
  Postoperative hospital（days）stay after lung transplantation
In-hospital mortality | Collect data for an expected average about 2 hours
  The proportion of patients who died during the initial hospitalization period following lung transplantation surgery
30-day postoperative mortality | Collect data for an expected average about 2 hours
  Number of deaths within 30 days post-transplant) / (Total number of lung transplant recipients) × 100%；
90-day postoperative mortality | Collect data for an expected average about 2 hours
  Number of deaths within 90 days post-transplant) / (Total number of lung transplant recipients) × 100%
The duration of endotracheal intubation | Collect data for an expected average about 2 hours
  Duration of intubation should be recorded from surgery end-time to extubation

OTHER OUTCOMES:
Grade 3 Primary Graft Dysfunction (PGD) | Collect data for an expected average about 2 hours
  PGD3:A ratio of arterial oxygen partial pressure to fraction of inspired oxygen (PaO₂/FiO₂) < 200 mmHg with bilateral infiltrates on chest radiograph, or Requirement for extracorporeal life support (ECLS) within 72 hours postoperatively, or use of inhaled pulmonary vasodilators for >48 hours during mechanical ventilation.
Pulmonary Infection | Collect data for an expected average about 2 hours
  Radiologically confirmed by a staff radiologist as new or progressive pulmonary infiltrates on: Chest X-ray or Computed tomography (CT) scan
Acute Kidney Injury | Collect data for an expected average about 2 hours
  A rise in serum creatinine >120 μmol/L
Cardiovascular Events | Collect data for an expected average about 2 hours
  Acute myocardial infarction； heart failure；Cardiovascular hemorrhage；Clinically significant arrhythmias；Conduction system disorders；Cardiac arrest；Refractory hypotension due to cardiogenic sock.
Hepatic Dysfunction | Collect data for an expected average about 2 hours
  Aspartate aminotransferase (AST) >34 or Alanine aminotransferase (ALT) >40 U/L;
Cerebral Infarction | Collect data for an expected average about 2 hours
  Diagnosed by staff radiologists as new or progressive ischemic lesions on CT or MRI

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang 310000, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided